CLINICAL TRIAL: NCT01329952
Title: Reinfection Rates and Long Term Outcomes in Currently Injecting Drug Users Following Successful Treatment for Hepatitis C
Brief Title: Reinfection and Long Term Outcomes in Intravenous Drug Users (IVDUs) After Hepatitis C Treatment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Pennine Acute Hospitals NHS Trust (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Dr Joanne Baxter, North Manchester General Hospital, Delauneys Road, Crumpsall, Manchester, M8 5RB
Other Study IDs: HCV-NMGH
Record Dates: First submitted 2011-04-04; First posted 2011-04-06 (Estimated); Last update posted 2011-04-06 (Estimated); Status verified 2011-03

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples Without DNA — Blood will be taken for Hepatitis C RNA, plus Hepatitis C genotype if positive. Blood will also be taken for liver function tests and a full blood count.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Current intravenous drug users: Those who were actively injecting drugs at the time of their hepatitis C treatment.
- Past drug users: Those who stopped injecting drugs intravenously at least 6 months prior to the start of treatment for hepatitis C

SUMMARY:
The investigators will identify possible participants using our database of previously treated hepatitis c patients. The investigators will identify those who have documented evidence of current injecting drug use as a risk factor for acquisition of the virus. The investigators will then search for those who have received curative treatment between 2004-2010. This covers all patients in the current database. The investigators will include those over 18 years old. The investigators will exclude those patients who are coinfected with either hepatitis B or HIV. This is because both of these conditions can accelerate liver damage when in combination with hepatitis c.

The possible participants identified will be sent an information sheet giving a simple and clear outline of the proposed research. The investigator will try to obtain an au to date residential address from the PAS system in the NHS or through confirmation from the patients GP or drug worker. It will explain the purpose of the study, why they have been chosen, what taking part will involve, the potential advantages and disadvantages of taking part and that everything will be kept confidential. It will also outline who is conducting the study, how any expenses will be paid and contact details for any problems/complaints that arise.

Those interested in taking part will attend an appointment at the hospital after they have had the opportunity to read through the information leaflet. They will be given time to ask any questions they have about the study and have them answered fully. They will then be asked to sign two copies of a consent form in order to take their participation any further. Once this is complete they can have their first 'liver assessment'. The assessment will take approximately 30-45 minutes to complete.

The investigators will take three blood samples from them (approximately 10mls of blood or 4 teaspoons full). One sample is to measure the levels of hepatitis C virus in the blood. This will tell us whether there has been reinfection with hepatitis C. The second sample is to measure the levels of inflammation within the liver and the third sample is to measure the full blood count. The investigators will then perform a liver scan called a fibroscan. This is a noninvasive test similar to an ultrasound (that pregnant women have) and gives a reading that can tell us about any 'stiffness' in the liver. It takes approximately five to ten minutes to complete and involves the patient lying on their back with their right arm above their head for the duration of the scan. Following the scan the investigators will ask the participant to complete a short questionnaire. This will include questions about past and current drug use as well as any alcohol use. The answers will be kept strictly confidential. They will be stored in the researchers locked office and have no direct participant identifiers on them. They will simply have a study number on them.The participant will then be thanked for their time and offered £30 to cover all travel and time expenses for their visit.

They will be invited to attend for a further liver assessment one year after their first one and annually thereafter. This is optional and they are of course free to withdraw from the study at any time without needing to give a reason.

The investigators will be identifying participants at different points in time following their curative treatment. For example some will have been cured 5 year ago whereas other will have been cured 6-12 months ago. This will increase the number of patient years follow up. Once the investigators have done the first set of liver assessment the participants will then be followed prospectively for as long as they wish to participate.

For the purpose of my higher degree I will present the data I have following two years of 'liver assessments'.

DETAILED DESCRIPTION:
There is a stark paucity of data published concerning reinfection rates post successful treatment for HCV in currently injecting drug users. The investigators research will focus in this important area and provide desperately needed evidence to increase confidence in treating this population who carry the burden of the disease. Treating larger numbers of individuals in this population will reduce the incidence of HCV in injecting drug users and therefore reduce the overall prevalence of the disease. This will reduce the current threat to public health that HCV produces.

DETAILS OF MD RESEARCH PROJECT

STUDY HYPOTHESIS:

HCV therapy in the currently injecting group is beneficial with reinfection rates and long term outcomes comparable to those who are not current injectors.

AIMS:

1. The main aim is to determine if patients who have been successfully treated for HCV and who are currently injecting drug users have comparable rates of reinfection to those who injected drugs in the past (at least 6 months ago).
2. A secondary aim is to determine if currently injecting drug users have comparable long term outcomes to those who injected drugs in the past (at least 6 months prior to treatment) in terms of liver fibrosis and progression.

OBJECTIVES:

1. To determine the rates of reinfection in an historical cohort of drug users with HCV who have been previously treated and achieved SVR compared to those who have injected drugs in the past (at least 6 months prior to treatment) and achieved SVR with treatment.
2. To determine long term outcomes in those who injected drugs at the time of treatment and compare this to past injecting drug users (those who injected drugs at least 6 months prior to treatment).

RESEARCH QUESTIONS:

1. Do current drug users have higher rates of reinfection than past drug users?
2. Is the rate of reinfection in drug users as a whole low?
3. Does progression of fibrosis continue following successful treatment for HCV?
4. How often do currently injecting drug users stop injecting during or after treatment for HCV?
5. How often do past drug users return to injecting drug use during or following treatment?
6. Does any rise in liver enzymes persist following successful treatment?
7. What are the most commonly used drugs for injection?
8. How often do currently injecting drug users share needles/equipment?
9. Do injecting drug users know that they can be reinfected following SVR?
10. What proportion of injecting drug users drink more than the recommended weekly allowance for alcohol?
11. What is the quality of life post SVR?

METHODOLOGY

STUDY DESIGN:

This is a prospective study looking at reinfection rates based on a historical cohort of intravenous drug users that have been previously treated and achieved an SVR.

PARTICIPANTS:

There is a HCV database set up at North Manchester Hospital of all patients started on treatment since 2004. The investigator will access this and create a separate database of those patients with injecting drug use at any time as their risk factor for acquisition of HCV. The investigator will then identify those who were injecting drugs in the 6 months prior to treatment including those who continued to inject during treatment. These will be the 'active' drug using group. The investigator will then identify the group of patients that stopped injecting drugs at least 6 months prior to commencing treatment. These will be the 'past' drug using group.

CONSENT:

The investigator will be responsible for obtaining informed consent from the participants. Two copies of the consent form will be obtained - one for the participants records and one for the study file. Prior to obtaining informed consent The investigator will highlight that if any information comes to light during the course of the study pertaining to a potential criminal activity The investigator will obliged to pass this information on to the relevant authorities.

DATA COLLECTION:

All potential participants will be sent written information detailing the study and inviting them to take part. This is to avoid any possible selection bias. The investigators aim to follow up this group for 2 years to collect data on outcomes including reinfection rates using annual HCV RNA (with subsequent genotyping if positive) and liver disease progression using standard liver function blood tests and a fibroscan (a non-invasive method to assess liver fibrosis and cirrhosis).

A questionnaire regarding drug use post treatment will be done detailing any high risk practises. They will also be questioned again about drug use on treatment in order to confirm which group they should be assigned to and to reduce the possibility of previous underreporting for fears of exclusion from the treatment programme initially. Alcohol history will also be assessed. Quality of life questionnaires validated for use in HCV will be used during follow up.

The investigator is aiming to recruit 45 participants in to each group. The participants will be asked to attend for 2 visits in total one year apart. One major limitation of this study is the frequency of sampling for HCV RNA. By doing this annually the investigators may miss those reinfections that the patient clears spontaneously. However, the investigator feels that it is those with persistent viraemia and therefore persistent reinfection that are important to quantify. This is because much of the physicians' reluctance to treat active drug users comes from the perception that reinfection will occur resulting in the need for further repeated courses of treatment. Whilst those transient reinfections that the investigators may miss are very important in terms of onwards transmission, they largely do not result in the need for further treatment.

DATA HANDLING:

All new data gathered will be included in a specially designed database which will be password protected and on a limited access drive on the NHS computer, following the principles set out in the data protection act. Identifiers will be kept to an absolute minimum. Data will be stored for 25 years before being destroyed.

COMMUNICATION OF RESULTS:

The investigator is aiming to distribute and communicate the results of this study at national and international conferences. The investigator is also aiming to publish a paper in a peer reviewed journal. The participants will be informed prior to consenting that they are entitled to access to the overall results.

ELIGIBILITY:
Inclusion criteria

* Aged 18 years or older
* Achieved cure (negative Hepatitis C pcr 6 months after completing treatment)
* Previous history of injecting drug use
* Previously infected with Hepatitis C

Exclusion criteria

* Prison resident
* Co-infection with HIV or chronic hepatitis B
* Did not achieve cure with treatment for Hepatitis C
* Pregnant females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This will focus specifically on long term outcomes for patients who are current and past injecting drug users at the time of their treatment. Injecting drug users who have already completed therapy and achieved SVR will be asked to return for assessment. During this study, the investigators will also enquire about any drug use prior to, during and after completing therapy. The investigators will compare this group with past injectors, (last injected at least 6 months prior to starting treatment) a group that most centres would consider appropriate for treatment).
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2011-05; Primary Completion 2013-05 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
To determine the reinfection rates in a historical cohort of drug users with Hepatitis C genotype 3 who have been previously treated and cured. | 2 years
  This will be calculated in terms of cases per 100 person years.

SECONDARY OUTCOMES:
To determine long term outcomes in those who injected drugs at the time of treatment and compare this to past injecting drug users. | 2 years
  Blood taken for HCV RNA +/- HCV genotype, liver function tests and full blood count. Annual fibroscans will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne M Baxter, MBChB, Principal Investigator — North Manchester General Hospital
Locations (1):
- North Manchester General Hospital, Manchester, Greater Manchester, United Kingdom